CLINICAL TRIAL: NCT00667238
Title: Functional Impact of Chronic Pediatric Pain
Brief Title: Chronic Pediatric Pain
Status: Withdrawn | Type: Observational
Why Stopped: Study never started due to resource related challenges
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rashmi Parekh Bhandari, Clinical associate professor, Stanford University
Other Study IDs: SU-04082008-1086
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

INTERVENTIONS:
Behavioral: Questionnaire

SUMMARY:
The purpose will be to study the functional impact of pediatric chronic pain on children, and their families. Focus will be on the impact of pain on school functioning, social functioning, psychological functioning and family functioning of pediatric chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have completed parent surveys before coming to the multidisciplinary pain management clinic evaluations.

Exclusion Criteria:

* If the patient's surveys are missing or incomplete (i.e. more than half of the survey was not completed, they will be excluded from entry into the data base.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 8-18
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2008-11-01 (Estimated); Study Completion 2008-11-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Parekh Bhandari, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States